CLINICAL TRIAL: NCT00005646
Title: Phase II Trial of Weekly Dose-Dense Paclitaxel in Extensive Stage Small Cell Lung Cancer
Brief Title: Paclitaxel in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39901; U10CA031946 (NIH); CLB-39901; CDR0000067826 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-05-02; First posted 2003-12-17 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel (Experimental): Patients receive paclitaxel for up to 4 cycles. One cycle = weekly drug for 6 weeks and 2 weeks rest
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel — 150 mg/sq m IV over 3 hours weekly for 6 weeks per cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete and overall response rate to paclitaxel in patients with previously untreated extensive stage small cell lung cancer. II. Determine the overall and progression free survival of these patients in response to this treatment regimen. III. Determine the toxicity of this treatment regimen in this patient population.

OUTLINE: This is a multicenter study. Patients receive paclitaxel IV over 3 hours weekly for 6 consecutive weeks. Treatment continues every 8 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months for 1 year, then every 3 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed extensive stage small cell carcinoma of the bronchus Extrathoracic metastatic disease, malignant pleural effusion, bilateral or contralateral supraclavicular adenopathy or contralateral hilar adenopathy Measurable disease One lesion that measures at least 20 mm in diameter using conventional techniques or at least 10 mm with spiral CT scan Lesions not considered measurable include: Bone lesions Leptomeningeal disease Ascites Pleural/pericardial effusion Cystic lesions Tumor lesions situated in a previously irradiated area Abdominal masses not confirmed and followed by imaging techniques No disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal, and/or ipsilateral supraclavicular nodes

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CTC 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT less than 2 times upper limit of normal Bilirubin less than 1.5 mg/dL Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No concurrent hormonal therapy except steroids for renal failure or hormones administered for nondisease related conditions Radiotherapy: At least two weeks since prior radiotherapy No concurrent palliative radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-04; Primary Completion 2004-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Response Rate | 1 year post treatment

SECONDARY OUTCOMES:
Progression-free survival | 12 months post treatment
Overall survival | 12 months post treatment
Overall response | 12 months
Toxicity | 1 year post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Socinski, MD, Study Chair — University of North Carolina
Locations (5):
- United States (5):
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Background] Blackstock AW, Herndon JE 2nd, Paskett ED, Miller AA, Lathan C, Niell HB, Socinski MA, Vokes EE, Green MR; Cancer and Leukemia Group B. Similar outcomes between African American and non-African American patients with extensive-stage small-cell lung carcinoma: report from the Cancer and Leukemia Group B. J Clin Oncol. 2006 Jan 20;24(3):407-12. doi: 10.1200/JCO.2005.02.1436. Epub 2005 Dec 19. PMID 16365181
- [Result] Graziano SL, Herndon JE 2nd, Socinski MA, Wang X, Watson D, Vokes E, Green MR; Cancer and Leukemia Group B. Phase II trial of weekly dose-dense paclitaxel in extensive-stage small cell lung cancer: cancer and leukemia group B study 39901. J Thorac Oncol. 2008 Feb;3(2):158-62. doi: 10.1097/JTO.0b013e318161225e. PMID 18303437
- [Result] Graziano SL, Socinski MA, Herndon JE, et al.: Dose-dense weekly paclitaxel (P) in extensive stage small cell lung cancer (ES-SCLC): Cancer and Leukemia Group B (CALGB) 39901. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2598, 646, 2003.